CLINICAL TRIAL: NCT03943615
Title: An Open-Label, Expanded Access Protocol for Patients With Sickle Cell Disease Who Have No Alternative Treatment Options
Brief Title: Expanded Access to Voxelotor for Patients With Sickle Cell Disease Who Have No Alternative Treatment Options
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: GBT440-037; C5341044 (Other: Alias Study Number)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Voxelotor
  Other Names: GBT440

SUMMARY:
The intent of this open-label, multicenter expanded access program (EAP) is to provide early access to voxelotor prior to market authorization

DETAILED DESCRIPTION:
The purpose of this program is to provide early access to voxelotor for patients with sickle cell disease who have exhausted alternative treatment options and are ineligible for actively-recruiting clinical trials of voxelotor.

This EAP may continue until such time that voxelotor is commercially available or the Sponsor discontinues the voxelotor EAP. Discontinuation may occur earlier if an individual participant or physician or Sponsor Medical Monitor decides to discontinue treatment.

ELIGIBILITY:
Inclusion Criteria

1. Documented diagnosis of sickle cell disease of any genotype confirmed by laboratory testing during screening
2. Ineligible or unable to participate in actively recruiting clinical studies of voxelotor
3. Hemoglobin (Hb) ≤ 10.5 g/dL during screening
4. No alternative treatment options in the judgment of the treating investigator
5. Participants, who if female and of child bearing potential, agree to use highly effective methods of contraception from study start to 30 days after the last dose of voxelotor, and who if male, agree to use barrier methods of contraception from study start to 30 days after the last dose of voxelotor
6. Patient has provided documented informed consent (the informed consent form [ICF] must be reviewed and signed by each participant),or for participants under 18 years of age, signed parental/legal guardian consent and participant assent.

Exclusion Criteria

1. Female who is breast feeding or pregnant
2. Hepatic dysfunction characterized by alanine aminotransferase (ALT) >4 × ULN
3. Patients with clinically significant bacterial, fungal, parasitic, or viral infection which require therapy:

   * Patients with acute bacterial infection requiring antibiotic use should delay screening/enrollment until the course of antibiotic therapy has been completed.
   * Patients with known active hepatitis A, B, or C or who are known to be human immunodeficiency virus (HIV) positive
4. Renal dialysis
5. Non-SCD conditions or complications of SCD for which survival beyond 3 months is unlikely, in the opinion of the treating Investigator
6. Any condition affecting drug absorption, such as major surgery involving the stomach or small intestine (prior cholecystectomy is acceptable)
7. Participated in another clinical trial of an investigational agent (or medical device) within 30 days or 5 half-lives of date of informed consent, whichever is longer, or is currently participating in another trial of an investigational agent (or medical device)
8. Medical, psychological, or behavioral conditions, which, in the opinion of the Investigator, may preclude safe participation, interfere with compliance or preclude informed consent

The Sponsor Medical Monitor makes the sole and final enrollment determination for any patient.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - Alabama Oncology, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - The John Hopkins Hospital, Baltimore, Maryland
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Queens Hospital Center, Jamaica, New York
  - Montefiore Medical Center PRIME, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Department of Pediatrics, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - VCU Health, Richmond, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-037